CLINICAL TRIAL: NCT06545500
Title: A Phase IIb, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy, Safety, and Pharmacokinetics of Glycopyrrolate Inhalation Solution Over 1 Week in Subjects With COPD
Brief Title: A Phase IIb Study of Glycopyrrolate Inhalation Solution Over 1 Week in Subjects With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-CO-211
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: Each participant is expected to complete all 4 treatment periods, each consisting of a different dose level of blinded medication depending on the treatment sequence they were assigned to
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level A (Experimental): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Interventions: Drug: Glycopyrrolate (85 μg)
- Dose Level B (Experimental): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Interventions: Drug: Glycopyrrolate (42.5 μg)
- Dose Level C (Experimental): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Interventions: Drug: Glycopyrrolate (14 μg)
- Dose Level D (Placebo Comparator): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glycopyrrolate (85 μg) — Administered by a standard jet nebulizer, twice daily for 7 consecutive days
  Arms: Dose Level A
Drug: Glycopyrrolate (42.5 μg) — Administered by a standard jet nebulizer, twice daily for 7 consecutive days
  Arms: Dose Level B
Drug: Glycopyrrolate (14 μg) — Administered by a standard jet nebulizer, twice daily for 7 consecutive days
  Arms: Dose Level C
Drug: Placebo — Administered by a standard jet nebulizer, twice daily for 7 consecutive days
  Arms: Dose Level D

SUMMARY:
This study is a randomized, double-blind, placebo-controlled complete block cross-over study designed to assess the efficacy, safety, and pharmacokinetics of 3 dose levels of glycopyrrolate inhalation solution delivered twice daily via standard jet nebulizer over three 1-week active treatment periods and one 1-week placebo period in subjects with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
Participants enrolled will be expected to participate for approximately 10 weeks;1-2 weeks for screening, four 1-week treatment periods separated by 1 week of washout between each treatment, and 1 week of follow-up. Participants will be randomized to a treatment sequence, 1-4, which will determine the order that they receive the dose levels during the four treatment periods of the study. Neither participants nor study staff will know which dose a participant is receiving in any given treatment period. All participants will receive all 4 dose levels and it is expected that each participant completes all four treatment periods in their assigned sequence. The primary objective of this study is to evaluate the bronchodilator effect of twice daily inhaled glycopyrrolate solution over a dose range administered by standard jet nebulizer in subjects with COPD on Day 7, to support the selection of the glycopyrrolate doses for further clinical development in a fixed-dose combination with ensifentrine.

ELIGIBILITY:
Inclusion Criteria:

* Males are eligible to participate if they agree to use contraception from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication.
* Females are eligible to participate if they are not pregnant, not breastfeeding, and ≥ 1 of the following conditions apply:

  1. Not a woman of childbearing potential (WOCBP) OR
  2. A WOCBP who agrees to follow the contraceptive guidance from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication.
* Current or former cigarette smokers with a history of cigarette smoking ≥ 10 pack years at Screening [number of pack years = (number of cigarettes per day / 20) × number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Pipe and/or cigar use cannot be used to calculate pack-year history. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Screening. Smoking cessation programs are permitted during the study.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines with symptoms compatible with COPD.
* Post-bronchodilator (4 puffs of salbutamol) spirometry at Screening demonstrating both the following:

  1. FEV1/forced vital capacity (FVC) ratio of < 0.70 AND
  2. FEV1 ≥ 30 % and ≤ 70% of predicted normal
* A posterior-anterior chest x-ray (CXR) at Screening or within 12 months prior to Screening showing no clinically significant abnormalities unrelated to COPD. If a CXR within the past 12 months is not available but a computed tomography (CT) scan within the same time period is available, the CT scan may be reviewed in place of a CXR.
* Capable of withdrawing from short-acting bronchodilators for 4 hours prior to spirometry testing and from BID LABA ± ICS therapy for 24 hours prior to spirometry.
* Capable of using the study nebulizer correctly.
* Ability to perform acceptable spirometry in accordance with ATS/ERS guidelines
* Willing and able to attend all study visits and adhere to all study assessments and procedures.

Exclusion Criteria:

* Concomitant clinically significant pulmonary disease other than COPD (i.e., asthma, tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnea (unless controlled with stable continuous positive airway pressure [CPAP] use), known alpha-1 antitrypsin deficiency, core pulmonale or other non-specific pulmonary disease).
* Within 6 months prior to Screening:

  1. COPD exacerbation requiring hospitalization.
  2. Use of therapies for COPD exacerbation (e.g., oral, intravenous, or intramuscular glucocorticoids).
* Lower respiratory tract infection within 6 weeks of Screening or an active infection at Screening.
* History of life-threatening COPD, including Intensive Care Unit admission and/or requiring intubation.
* Previous lung resection or lung reduction surgery within 1-year of Screening.
* Long term oxygen use defined as oxygen therapy prescribed for greater than 12 hours per day. As needed oxygen use (≤ 12 hours per day) is not exclusionary.
* Severe comorbidities including unstable cardiac, or any other clinically significant medical conditions including uncontrolled diseases that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject.
* History of or clinically significant on-going bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within the previous 6 months.
* History of narrow angle glaucoma.
* History of hypersensitivity or intolerance to aerosol medications, salbutamol or glycopyrrolate or any of its excipients/components, anticholinergic agents, or sympathomimetic amines.
* Pulmonary rehabilitation unless such treatment has been stable from 4 weeks prior to Screening (Visit 1) and remains stable during the study. Pulmonary rehabilitation programs should not be started or completed during participation in the study.
* Major surgery (requiring general anesthesia) in the 6 weeks prior to Screening, lack of full recovery from surgery at Screening, or planned surgery through the end of the study.
* History of or current malignancy of any organ system, treated or untreated within the past 5 years, except for localized basal or squamous cell carcinoma of the skin.
* Current or history of drug or alcohol abuse within the past 5 years.
* Estimated glomerular filtration rate (eGFR) < 30 mL/min.
* Women who are breast feeding.
* Use of an experimental drug within 30 days or within 5 half-lives of Screening, whichever is longer, and/or participation in a study treatment-free follow-up phase of a clinical study within 30 days prior to Screening.
* Use of an experimental medical device or participation in a follow-up phase of an experimental medical device clinical study within 30 days prior to Screening.
* Affiliation with the investigator site, including an Investigator, Sub-Investigator, study coordinator, study nurse, other employee of participating investigator or study site or a family member of the aforementioned.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-01-02 (Actual); Study Completion 2025-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Clinical Research of West Florida Inc - Tampa, Tampa, Florida
  - Midwest Chest Consultants PC, Saint Charles, Missouri
  - American Health Research Inc, Charlotte, North Carolina
  - Velocity Clinical Research - Greenville, Greenville, South Carolina
  - Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - Velocity Clinical Research - Union, Union, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Demographic and baseline characteristics are presented by sequence assignment based on which treatment sequence the participant was randomized to. Each treatment sequence was comprised of four treatment periods with a different dose level being received during each period. Therefore, each participant received each dose and there is no demographic or baseline data based dose alone.
Groups:
- Sequence 1: Participants assigned to treatment Sequence 1 received dose level A for treatment period 1, followed by dose level D for treatment period 2, then dose level B for treatment period 3, and finished with dose level C for treatment period 4
- Sequence 2: Participants assigned to treatment Sequence 2 received dose level B for treatment period 1, followed by dose level A for treatment period 2, then dose level C for treatment period 3, and finished with dose level D for treatment period 4
- Sequence 3: Participants assigned to treatment Sequence 3 received dose level C for treatment period 1, followed by dose level B for treatment period 2, then dose level D for treatment period 3, and finished with dose level A for treatment period 4
- Sequence 4: Participants assigned to treatment Sequence 4 received dose level D for treatment period 1, followed by dose level C for treatment period 2, then dose level A for treatment period 3, and finished with dose level B for treatment period 4
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 11 | 12 | 11
Completed | 10 | 11 | 11 | 9
Not Completed | 2 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Not Wanting Further Contact | 1 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 1 | 0 | 0 | 0
Not completed — Withdrawal Due to Hurricane | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 12 | 11 | 12 | 11 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (7.15) | 68.7 (4.54) | 62.5 (9.17) | 66.1 (6.28) | 65.1 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 7 | 7 | 28
  Male | 4 | 5 | 5 | 4 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 9 | 12 | 10 | 40
  Black | 3 | 2 | 0 | 1 | 6
  Asian | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0
  Multiple | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  HISPANIC OR LATINO | 1 | 0 | 0 | 0 | 1
  NOT HISPANIC OR LATINO | 10 | 11 | 12 | 9 | 42
  NOT REPORTED | 1 | 0 | 0 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 12 | 11 | 46
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.68 (6.284) | 29.04 (2.363) | 28.98 (9.098) | 27.55 (4.473) | 28.83 (6.016)
Childbearing potential [Count of Participants; unit: Participants] — Population: Demographic is specific to female population only
  Participants
    Yes: number analyzed (Participants) | 8 | 6 | 7 | 7 | 28
    Yes | 0 | 0 | 0 | 0 | 0
    No: number analyzed (Participants) | 8 | 6 | 7 | 7 | 28
    No | 8 | 6 | 7 | 7 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Average Baseline in Morning Trough Forced Expiratory Volume in 1 Second (FEV1)
Time Frame: Baseline (pre-dose for each treatment period) and Day 7
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Dose Level A Glycopyrrolate (85 μg): The treatment period was 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Glycopyrrolate (85 μg): Administered by a standard jet nebulizer, twice daily for 7 consecutive days
- Dose Level B Glycopyrrolate (42.5 μg): The treatment period was 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Glycopyrrolate (42.5 μg): Administered by a standard jet nebulizer, twice daily for 7 consecutive days
- Dose Level C Glycopyrrolate (14 μg): The treatment period was 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Glycopyrrolate (14 μg): Administered by a standard jet nebulizer, twice daily for 7 consecutive days
- Dose Level D (Placebo): The treatment period was 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Placebo: Administered by a standard jet nebulizer, twice daily for 7 consecutive days
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.0525 (0.02125) | 0.0393 (0.02135) | 0.0115 (0.02069) | -0.0287 (0.02029)

2. Secondary Outcome: Change From Average Baseline FEV1 to Average Peak FEV1 Measured Over 4 Hours
Time Frame: Baseline (pre-dose for each treatment period) and Day 7
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.2333 (0.02304) | 0.2042 (0.02314) | 0.1568 (0.02243) | 0.0520 (0.02200)

3. Secondary Outcome: Change From Average Baseline FEV1 to Average FEV1 Area Under the Curve Versus Time From Time 0 to 4 Hours (AUC0-4h)
Description: The endpoint is measured as AUC/4 hour time interval resulting in an average volume measure in liters.
Time Frame: Baseline (pre-dose for each treatment period) and Day 7
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.0969 (0.02037) | 0.0693 (0.02046) | 0.0418 (0.01984) | -0.0403 (0.01945)

4. Secondary Outcome: Change From Average Baseline FEV1 to Average FEV1 Area Under the Curve Versus Time From Time 0 to 12 Hours (AUC0-12h)
Description: The endpoint is measured as AUC/12 hour time interval resulting in an average volume measure in liters.
Time Frame: Baseline (pre-dose for each treatment period) and Day 7
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.0916 (0.02006) | 0.0656 (0.02031) | 0.0338 (0.02039) | -0.0449 (0.01927)

5. Secondary Outcome: Change From Average Baseline FEV1 to Evening Trough FEV1
Time Frame: Baseline (pre-dose for each treatment period) and Day 7
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.0652 (0.02054) | 0.0569 (0.02066) | 0.0091 (0.02115) | -0.0484 (0.01996)

6. Secondary Outcome: Change From Average Baseline FEV1 to Peak FEV1 Measured Over 4 Hours After First Dose
Time Frame: Baseline (pre-dose) and Day 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.2117 (0.01786) | 0.1872 (0.01798) | 0.1643 (0.01675) | 0.0730 (0.01716)

7. Secondary Outcome: Change From Average Baseline FEV1 to Average FEV1 AUC0-4h Measured After First Dose
Description: The endpoint is measured as AUC/4 hour time interval resulting in an average volume measure in liters.
Time Frame: Baseline (pre-dose) and Day 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 39 | 40 | 41 | 40
Liters | 0.1377 (0.01498) | 0.1027 (0.01507) | 0.0859 (0.01405) | 0.0000 (0.01439)

8. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Time Frame: From first dose through the follow-up contact (approximately 8 weeks per participant). Overall safety data was collected for 5 months total.
Measure: Number; unit: Events
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
Number analyzed (Participants) | 40 | 40 | 41 | 43
Events | 13 | 8 | 7 | 15

9. Secondary Outcome: Glycopyrronium Free Base AUC0-12h
Time Frame: After morning dose Day 7
Population: Placebo was excluded from the PK concentration listings.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg)
Number analyzed (Participants) | 22 | 22 | 19
h*pg/mL | 256 (187.7) | 108 (66.22) | 38.4 (18.25)

10. Secondary Outcome: Glycopyrronium Free Base Maximum Plasma Drug Concentration (Cmax)
Time Frame: After morning dose Day 7
Population: Placebo was excluded from the PK concentration listings.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg)
Number analyzed (Participants) | 22 | 22 | 19
pg/mL | 53.7 (38.46) | 24.7 (13.87) | 9.27 (5.354)

11. Secondary Outcome: Glycopyrronium Free Base Time to Maximum Plasma Drug Concentration (Tmax)
Time Frame: After morning dose Day 7
Population: Placebo was excluded from the PK concentration listings.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg)
Number analyzed (Participants) | 22 | 22 | 19
hours | 0.33 [0 to 1.63] | 0.33 [0 to 0.77] | 0.43 [0.25 to 1.25]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 5-month period, however individual participant data was collected only for 8 weeks
Description: Adverse events are assessed at every participant visit and end of study follow up call
Groups:
- Dose Level A Glycopyrrolate (85 μg): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Glycopyrrolate (85 μg): Administered by a standard jet nebulizer, twice daily for 7 consecutive days
- Dose Level B Glycopyrrolate (42.5 μg): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Glycopyrrolate (42.5 μg): Administered by a standard jet nebulizer, twice daily for 7 consecutive days
- Dose Level C Glycopyrrolate (14 μg): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Glycopyrrolate (14 μg): Administered by a standard jet nebulizer, twice daily for 7 consecutive days
- Dose Level D (Placebo): The treatment period will be 7 days, followed by a 7-day washout period, before beginning the next treatment in the sequence they were assigned to
  Placebo: Administered by a standard jet nebulizer, twice daily for 7 consecutive days
Arm/Group | Dose Level A Glycopyrrolate (85 μg) | Dose Level B Glycopyrrolate (42.5 μg) | Dose Level C Glycopyrrolate (14 μg) | Dose Level D (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 2/40 | 1/40 | 0/41 | 1/43
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/41 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level A Glycopyrrolate (85 μg) (N=40) | Dose Level B Glycopyrrolate (42.5 μg) (N=40) | Dose Level C Glycopyrrolate (14 μg) (N=41) | Dose Level D (Placebo) (N=43)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0 | 0
INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-10-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT06545500/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT06545500/SAP_001.pdf